CLINICAL TRIAL: NCT06222242
Title: mychoiceTM Implementation in a Real World Clinical Environment - Delivery and Effectiveness
Brief Title: mychoiceTM Implementation With Medical Oncology Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Linda Fleisher, Research Professor, Fox Chase Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-8003
Record Dates: First submitted 2023-12-08; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mychoiceTM intervention (Experimental): Single arm study - all participants receive mychoiceTM
  Interventions: Behavioral: mychoiceTM

INTERVENTIONS:
Behavioral: mychoiceTM — mychoiceTM is an online, educational tool designed to help prepare patients for a conversation with their provider about clinical trials as a treatment option. It consists of text, animations, and videos of real cancer patients sharing their experience with clinical trials. It is not meant to be a recruitment tool, but rather a preparatory tool to promote shared decision making between patients and providers.

SUMMARY:
This is a pragmatic, non-randomized mixed-methods evaluation study designed to evaluate the feasibility and acceptability of delivering the mychoiceTM tool to new Medical Oncology patients as well as to more deeply explore its value to patients in their discussion with their provider about clinical trials as a treatment option over the course of their oncology treatment (Effectiveness).

DETAILED DESCRIPTION:
This is a pragmatic, non-randomized mixed-methods evaluation study designed to evaluate the feasibility and acceptability of delivering the mychoiceTM tool to new Medical Oncology patients as well as to more deeply explore its value to patient in their discussion with their provider about clinical trials as a treatment option over the course of their oncology treatment (Effectiveness).

Our goal is to focus this study with patients who have had their first Medical Oncology Appointment based on a nightly EMR feed. The mychoiceTM link (currently mychoice.kevindurr.com, but will change to mychoice.templehealth.org prior to study launch) will be sent to patients through a REDCap feed where they can review the mychoice tool and voluntarily answer a short 5 question quality improvement (QI) survey about their experience with mychoiceTM. The survey will include a question about their willingness to be contacted regarding the more in-depth effectiveness study. This survey data will only be evaluated at an aggregate level and used for process improvement purposes.

The effectiveness study will be conducted with patients who have used mychoiceTM and have agreed to be contacted by Fox Chase Research Staff as indicated in their response to one of the questions in the QI survey. Our goal is to conduct follow-up with those patients who used mychoiceTM to evaluate the impact of the tool on patients' perceived preparedness to discuss clinical trials with their physician and insights into this decision-making process over six-months during their treatment. In addition, we will assess provider and system barriers and facilitators to implementation of mychoice in real world settings to guide future dissemination and implementation.

There are three levels of evaluation questions in this project and specific aims related to each.

1. Can an evidence-based digital health tool designed to promote discussion about clinical trial participation (mychoiceTM) be easily provided to patients in real time, and will this dissemination approach be acceptable to patients and providers? (Aim 1)
2. For a sub-set of these patients who use the tool and express interest in participating in a follow-up study evaluation, does the tool positively impact their preparation for a discussion about clinical trials participation across their cancer treatment trajectory? (Aim 3. What are the factors (based on Implementation Research frameworks - RE-AIM and Consolidated Framework Implementation Research) that influence the implementation of mychoiceTM in a real world setting that can guide future dissemination and implementation.

Therefore, the aims of this pragmatic, non-randomized, mixed-methods study is to assess the feasibility, acceptability (Aim 1) and effectiveness of the mychoiceTM preparatory tool for patients (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

18 years of age or over

Able to speak and read English

Medical Oncology patients who have had their initial visit

Have a cell phone number and/or an email in the electronic medical record

Exclusion Criteria

Doesn't not speak or read English

Patients who do not have a cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility to disseminate the mychoice tool to patients | 24 months
  Assess the feasibility of disseminating the mychoiceTM preparatory tool to all Medical Oncology patients and the acceptability (measured by recommendation to other patients. Patient feasibility will focus on the proportion of patients who receive the mychoiceTM tool and open the web-based intervention (goal 50%).
Acceptability | 24
  Patient acceptability will be measured for those patients who complete a voluntary, anonymous, feedback survey. Patients will rate how much they would recommend the navigation intervention to other patients on a scale of 1 to 5. Acceptability threshold would be met with a mean score of 3.5 or higher across all patients (aggregated data) who complete the feedback form (QI).
Effectiveness | 24 months
  Assess the effectiveness and value of the mychoiceTM tool on patients' preparation for the discussion about clinical trials through baseline and 4 monthsurveys and interviews with a selected sample at 2 months. The primary outcome will be to measure the effectiveness of the tool using a modified Ottawa Preparation Scale (PrepDM, 1-5 scale) addressing the effectiveness of the tool to prepare for a discussion with their provider. Based on our previous randomized trial, benchmark for success is mean score of 3.5 or higher across all patients enrolled on the PrepDM measures (or a total score of 62.5).

SECONDARY OUTCOMES:
Implementation Factors | 24 months
  We will assess implementation factors (both barriers and facilitators) at the provider and institutional levels, through review of implementation notes from planning and implementation meetings, as well as study notes using a coding form based on the domains of the Consolidated Framework for Implementation Research and distribute post-launch provider surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Fleisher, PhD, MPH, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States